CLINICAL TRIAL: NCT01126463
Title: Phase 1 Study of Hepatic Intra-Arterial Administration of 188RE-SSS Lipiodol to Treat HepatoCellular Carcinomas
Brief Title: 188RE-SSS Lipiodol to Treat HepatoCellular Carcinomas
Acronym: LIP-RE-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIP-RE-I
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinomas
Keywords: Hepatocellular carcinomas; lipiodol; rhenium; Non operable Hepatocellular carcinomas
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — rhenium-SSS-lipiodol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rhenium Lipiodol (Experimental): Hepatic Intra-Arterial Administration of radio-active lipiodol.
  Interventions: Drug: 188Re-SSS Lipiodol

INTERVENTIONS:
Drug: 188Re-SSS Lipiodol — Hepatic Intra-Arterial Administration of radio-active lipiodol.

SUMMARY:
This study is to determine the maximum tolerated dose and the recommended 188Re-SSS Lipiodol activity for hepatic intra-arterial injection in patients with hepato-cellular carcinoma. The new radioactive isotope 188Rhenium associated with Lipiodol is expected to reduce the radioprotection constraints and hence the duration of the hospitalisation in a protected room from 8 to 1 day.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most prevalent primary cancers in many countries. In France, mortality due to HCC on viral C cirrhosis is going to increase of about 150% for men and 200% for women until 2020. Consequently, HCC is a problem of public health.

The current treatment for HCC is mainly palliative with chemoembolization or intra-arterial radiotherapy, and intra-arterial targeted radiotherapy being the best tolerated method (iodine-131-labelled lipiodol being the most commonly used).

However, since 2007, a new therapeutic approach can be considered with oral sorafenib, an anti-angiogenic drug which increases slightly the survival of patients.

The key for an efficient treatment of HCC is presumably a co-treatment of sorafenib and intra-arterial radiotherapy. The 131I-lipiodol is a good candidate but presents disadvantages: it requires hospitalization in a radionuclide therapy room for one week. Therefore, it is necessary to find new radioactive labellings for lipiodol. In this objective, 188Re-SSS lipiodol, a new radioactive labeled stable complex has been developed. It has a short half-life and a tiny amount of gamma radiation compared to 131I-lipiodol, so it allows to reduce hospitalization in a protected room from 8 days to only one day.

The aim of this study is to determine the Maximum Tolerated Dose and thus the recommended activity of 188Re-SSS lipiodol by intra-arterial injection in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18,
* WHO performance status ≤ 2,
* Hepatocellular carcinoma histologically or cytologically proven, or association of liver tumor with chronic hepatopathy and AFP > 400 ng/ml, or tumorous hepatic formation considered as hypervascularised by at least 2 methods of imaging in cirrhotic patient, Non operable, non resectable, non transplantable, non accessible to percutaneous treatment tumor,
* Measurable tumor, uni- or multinodular, taking up less than 50% of hepatic volume,
* Stage A to C of the BCLC classification (or stage 0 to 4 of the CLIP) with:

  * No thrombosis of the portal vein, therapeutic escape or intolerance causing the end of the treatment or contraindication to sorafenib
  * If thrombosis of the portal vein, therapeutic escape to Lipiocis,
* Possibility of treatment by intra-arterial radiotherapy over a decision of a Multidisciplinary Committee,
* Written informed consent

Exclusion Criteria:

* Patient with a stage ≥ 3 toxicity of the CTCAE version 4
* Stage D of the classification BCLC
* Acute impairment of hepatic functions (Child-Pugh B9 or C)
* Grade III Hepatocarcinoma of the Okuda classification
* Encephalopathy with troubles even moderated of cognitive functions
* Advanced chronic respiratory insufficiency
* Creatinine clearance < 55 ml/min, polynuclear neutrophils < 1500 G/L, platelets < 50 G/L, prothrombin < 40% (INR > 2,3)
* Contraindication to the intra-arterial administration
* Patients who can't be followed up for psychological or geographic reasons
* Patients dependant on another person for daily care
* Urinary incontinence
* Progressive cancer
* Pregnant or breastfeeding woman, or not using adequate effective contraception method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose | Injection each week during 4 weeks and at month 2
  Toxicity CTC grade ≥ 3 with CTCAE version 4.

SECONDARY OUTCOMES:
Bio-availability | 1, 6, 24 et 48 hours after treatment injection
  Measurement by gamma-scintigraphy and by measurement of radio-activity in urinary, faecal and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne GARIN, MD, PhD, Principal Investigator — Centre Eugene Marquis
Locations (1):
- Centre Eugene Marquis, Rennes, France

REFERENCES:
- [Background] Garin E, Rakotonirina H, Lejeune F, Denizot B, Roux J, Noiret N, Mesbah H, Herry JY, Bourguet P, Lejeune JJ. Effect of a 188 Re-SSS lipiodol/131I-lipiodol mixture, 188 Re-SSS lipiodol alone or 131I-lipiodol alone on the survival of rats with hepatocellular carcinoma. Nucl Med Commun. 2006 Apr;27(4):363-9. doi: 10.1097/00006231-200604000-00008. PMID 16531923